CLINICAL TRIAL: NCT03185104
Title: Randomized Double-blind Placebo-controlled Trial of Silver Diamine Fluoride for Caries Prevention in Removable Partial Dentures Wearers
Brief Title: Silver Diamine Fluoride for Caries Prevention in Removable Partial Dentures Wearers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SDF RPD wearers
Record Dates: First submitted 2017-04-24; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Dental Caries; Dental Caries of Root Surface
Keywords: removable partial denture; silver diamine fluoride
MeSH Terms: conditions — Dental Caries; Root Caries | interventions — silver diamine fluoride

STUDY DESIGN:
Intervention Model Description: Removable partial denture wearers are randomized assigned to either the fluoride group or the placebo group. The fluoride group receives semi-annually professionally applied 38% SDF solution to all exposed tooth and root surfaces while the placebo group receives distilled water using the same application method.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Application of the SDF/placebo is conducted by a dentist who is not involved in the clinical data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silver diamine fluoride (Experimental): 38% silver diamine fluoride solution (Saforide, Toyo Seiyaku Kasei Co. Ltd., Osaka, Japan) is professionally applied to exposed coronal and root surfaces of all teeth every 6 months for 36 months.
  Interventions: Drug: Silver Diamine Fluoride
- Distilled water (Placebo Comparator): Distilled water is professionally applied to exposed coronal and root surfaces of all teeth every 6 months for 36 months.
  Interventions: Drug: Distilled Water

INTERVENTIONS:
Drug: Silver Diamine Fluoride — Silver diamine fluoride solution is applied to the dried and exposed coronal and root surfaces of all teeth by means of a disposable microbrush.
  Other Names: Saforide
  Arms: Silver diamine fluoride
Drug: Distilled Water — Distilled water is applied to the dried and exposed coronal and root surfaces of all teeth by means of a disposable microbrush.
  Arms: Distilled water

SUMMARY:
This study measures and compares the effect of silver diamine fluoride (SDF) on caries increment in removable partial denture wearers. Half of the participants will SDF and while the other half will receive placebo.

DETAILED DESCRIPTION:
Removable partial dentures are commonly constructed to replace missing teeth. It is observed that removable partial denture wearers are susceptible to dental caries.

The mode of action of silver diamine fluoride on caries prevention is dual: fluoride ions interact synergistically with silver to react with hydroxyapatite to form fluorapatite, and silver is bactericidal by reacting with the thiol groups of the amino and nucleic acids that halt the metabolic and reproductive functions of the cariogenic bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are wearing removable partial dentures constructed by staff or students at the Prince Philip Dental Hospital are recruited

Exclusion Criteria:

* If they have less than 4 teeth in any dental arch, have advanced periodontal disease in 2 or more sextants, have received therapeutic radiation of the head and neck region, have concurrent systemic illness that alters salivary flow, or have participated in a clinical trial within 6 months before the commencement of participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Caries increment | 36 months
  New and recurrent caries lesions are recorded according to the International Caries Detection and Assessment System (ICDAS). Molars and premolars are considered to have 5 coronal surfaces, whereas canines and incisors are considered to have 4. The cleaned and dried teeth are recorded as sound, sealed, restored, crowned, or missing. Each coronal tooth surface is classified using a 7-point ordinal scale ranging from sound to extensive cavitation using a WHO probe. The same procedure is repeated for all root surfaces. Coronal and root surface caries increments are calculated by comparing the baseline and follow-up observations for each tooth surface.

SECONDARY OUTCOMES:
Prevalence of oral colonization of oral yeasts | 36 months
  The prevalence of oral yeast in oral rinse and dental plaque is counted. Prevalence is expressed as percentage of the participants.
Colonization of oral yeasts in oral rinse | 36 months
  The count of oral yeasts in oral rinse is recorded. The count of oral yeast in oral rinse is expressed as colony-forming unit (cfu)/ml.
Colonization of oral yeasts in dental plaque | 36 months
  The count of oral yeasts in dental plaque is recorded. The count of oral yeast in dental plaque is expressed as cfu/g.
Prevalence of oral colonization of Streptococcus mutans (S. mutans) | 36 months
  The prevalence S. mutans in stimulated whole saliva (SWS) and dental plaque is counted. Prevalence is expressed as percentage of the participants.
Colonization of S. mutans in saliva | 36 months
  The count of S. mutans in SWS is recorded. The count of S. mutans in SWS is expressed as cfu/ml.
Colonization of S. mutans in dental plaque | 36 months
  The count of S. mutans dental plaque is recorded. The count of S. mutans in dental plaque is expressed as cfu/g.
Prevalence of oral colonization of lactobacilli | 36 months
  The prevalence of lactobacilli in SWS and dental plaque is counted. Prevalence is expressed as percentage of the participants.
Colonization of lactobacilli in saliva | 36 months
  The count of lactobacilli in SWS is recorded. The count of lactobacilli in SWS is expressed as cfu/ml.
Colonization of lactobacilli in dental plaque | 36 months
  The count of lactobacilli in dental plaque is recorded. The count of lactobacilli in dental plaque is expressed as cfu/g.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine CM Leung, BDS,MDS, PhD, Principal Investigator — Faculty of Dentistry, The University of Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided